CLINICAL TRIAL: NCT06906068
Title: Assessing the Impact of Probiotic Supplementation in Children Diagnosed With Autism Spectrum Disorder: the PROBI-O-TISM Study
Acronym: (PROBI-O-TISM)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valérie Marcil (Other)
Collaborators: Hôpital du Sacré-Coeur de Montréal (CIUSSS - NIM) (Unknown); University of Ottawa (Other); Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other); Institut National de la Recherche Scientifique - Centre Armand Frappier Santé Biotechnologie (Unknown)
Responsible Party: Sponsor-Investigator, Valérie Marcil, Professor, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2025-8319
Record Dates: First submitted 2025-03-19; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Gastrointestinal symptoms; Sleep disorder; Probiotics; Microbiota; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): A fermented probiotic beverage containing 3 lactobacilli
  Interventions: Dietary Supplement: Three strains of Lactobacillus: L. acidophilus CL1285®, L. casei LBC80R® and L. rhamnosus CLR2®
- Placebo (Placebo Comparator): A beverage without bacteria (identical taste and nutritional content to the probiotic beverage)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Three strains of Lactobacillus: L. acidophilus CL1285®, L. casei LBC80R® and L. rhamnosus CLR2® — A probiotic beverage (98 g) at dose of 50.10^9 CFU, taken once daily for 14 weeks.
  Arms: Probiotic
Other: Placebo — Non fermented beverage (98 g) with no probiotic strains, taken once daily for 14 weeks.
  Arms: Placebo

SUMMARY:
Children with autism spectrum disorder (ASD) present with stereotyped behaviors and often with comorbidities including gastrointestinal symptoms and sleep disturbances. These affect the quality of life of both children and parents. As of now, interventions available to manage ASD-related behaviors rely heavily on the services of professionals who are often difficult to access. What is even more striking is that there are currently no approved medications to treat the core symptoms of ASD. There is an important need for additional strategies to manage severity of ASD and to develop new treatments.

Targeting the bacteria living in the intestine, named 'gut microbiota', by using probiotics is an avenue that has been proposed by other groups to improve behaviors associated with ASD and gastrointestinal symptoms. However, these studies have important limitations, pressing the need for robustly designed interventions.

Previously, the PROBI-O-TISM pilot study was conducted at CHU Sainte-Justine. The investigators confirmed that the Bio-K+ probiotic beverage is acceptable and safe for autistic children and that the proposed study protocol is feasible. The study also led to promising preliminary results suggesting a beneficial effect of the probiotics on behaviors, gastrointestinal symptoms and sleep.

The proposed study will answer the question: ''Does supplementing with Bio-K+ probiotics reduce the severity of autistic behaviors and comorbidities in children with a diagnosis of ASD? '' The investigators will use a solid study design, a double-blinded randomized controlled-trial with placebo, to test the efficacy of a 14-week treatment with daily Bio-K+ probiotic supplement in children aged 4 to 11 years old. The investigators will also study the impact of the supplementation on other parameters such as quality of life, gut microbiota and brain signaling.

This is a unique opportunity to test a simple approach to improve behaviors and comorbidities in autistic children.

ELIGIBILITY:
Inclusion Criteria:

* Being an autistic child with normal intelligence as documented by a neuropsychology assessment at the time of ASD diagnosis based on the ADOS score and the clinical impression of a multidisciplinary team of experts in autism diagnosis in the Department of Psychiatry;
* Being between the ages of 4 and 11 years;
* Acceptance and ability of the child to consume the probiotics product.

Exclusion Criteria:

* Epilepsy;
* Autism in the context of a genetic syndrome such as Fragile X or Bourneville sclerosis;
* Known presence of cancer, diabetes, celiac disease or inflammatory bowel disease (Crohn's disease or ulcerative colitis);
* Genetic disorder such as trisomy 21 or 14;
* Immune system disorder;
* Intolerance or allergy to Bio-K+ pea-based probiotics;
* Having taken antibiotics or probiotics in the previous 3 months

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in ATEC (Autism Treatment Evaluation Checklist) total score between baseline and week 14 | 14 weeks
  Mean change in ATEC total score between baseline and week 14 will be compared to verify the supplementation effects. ATEC scale consists of 77 items grouped into four subscales: (1) language, (2) perception, (3) sociability and (4) behavior. The total score is 0-179; the higher the score, the more severe ASD-related behaviors

SECONDARY OUTCOMES:
Mean change in ATEC (Autism Treatment Evaluation Checklist) total score between week 14 and week 18 | 4 weeks
  Mean change in ATEC total score between week 14 and week 18 will be compared to verify persistence of treatment effects after wash-out (product cessation). The total score is 0-179; the higher the score, the more severe ASD-related behaviors.
Mean change in each ATEC (Autism Treatment Evaluation Checklist) sub-scores (language, perception, sociability, and behavior) between baseline , week 14 and week 18 . | Baseline, 14 weeks and 18 weeks
  Mean change in each ATEC sub-scores (language, perception, sociability, and behavior) will be compared between baseline, week 14 to verify supplementation effect and week 18 to evaluate persistence of treatment effects after wash-out (product cessation). The total score is 0-179; the higher the score, the more severe ASD-related behaviors.
Mean change in ATEC (Autism Treatment Evaluation Checklist) total score at week 4 and week 8 from baseline. | 4 weeks and 8 weeks
  Mean change in ATEC total score at week 4 and from baseline will be collected to document effect over time. The total score is 0-179; the higher the score, the more severe ASD-related behaviors
Mean change in VABS-III (adaptive behavior skills) total and sub-scores between baseline, week 14 and week 18. | Baseline, 14 weeks and 18 weeks
  Mean change in VABS-III total and sub-scores will be compared between baseline, week 14 to determine supplementation effect and week 18 to verify persistence of treatment effects after wash-out (product cessation). It consists of four subscales: communication, daily living skills, socialization and motor skills. The total score (range 0-72) and the four sub-scores total will be calculated. The higher scores indicate higher levels of functioning.
Mean change in 6-GSI (6-Gastrointestinal Severity Index) score between baseline, week 4, week 8, week 14 and week 18. | From baseline up to 18 weeks.
  Mean change in 6-GSI score will be compared between baseline, week 4, week 8, week 14 to evaluate supplémentation effect and week 18 to verify to persistence of treatment effects after wash-out (product cessation).The total score is 0-12, with higher values indicating greater severity.
Mean change in CSHQ (Child's Sleep Habits Questionnaire) total and sub-scores between baseline, week 4, week 8, week 14 and week 18. | From baseline up to 18 weeks
  Mean change in CSHQ total and sub-scores will be compared between baseline, week 4, week 8, week 14 to evaluate suplementation effects and week 18 to verify persistence of treatment effects after wash-out (product cessation). Total score is 33-99 divided in eight subscales: (1) bedtime resistance, (2) sleep-onset delay, (3) sleep duration, (4) sleep anxiety, (5) nocturnal awakenings, (6) parasomnias, (7) sleep disordered breathing and (8) morning waking/daytime sleepiness. The higher the CSHQ score the greater the complaints.
Mean change in Pediatric Quality of Life Inventory (PedsQL) score between baseline, week 14 and week 18. | Baseline, 14 weeks and 18 weeks
  Mean change in PedsQL score will be compared between baseline, week 14 to evaluate supplementation effects and week 18 to verify persistence of treatment effects after wash-out (product cessation). PedsQ consists in 23 items and four subscales: physical functioning, emotional functioning, social functioning and school functioning. A higher score represents better health related QoL.
Mean change in Parenting Stress Index-Short Form (PSI-SF) score between baseline, week 14 and week 18. | Baseline, 14 weeks and 18 weeks
  Mean change in PSI-SF score will be compared between baseline, week 14 to determine supplementation effects and week 18 to verify persistence of treatment effects after wash-out (product cessation). It is divided into three domains: parental distress, dysfunctional parent-child interaction and difficult child, with a total score ranging from 36 to 180. A higher score indicates a higher clinical level of distress.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Marcil, Professor, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
IPD might be shared to other research upon resonable request to the Principal Investigator/Sponsor.